CLINICAL TRIAL: NCT06615284
Title: A Phase 1 Randomized, Single-Blind, Three-Arm, Staggered Parallel Study to Assess the Safety, Tolerability, and Pharmacokinetics of Atorvo+™ in Healthy Adult Participants
Brief Title: A Study of Atorvo+™ in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indication Bioscience LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB.ATO-875
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Coronary Heart Disease; Dyslipidemias
Keywords: Atorvastatin; Cannabidiol; CBD; CHD; LDL-C
MeSH Terms: conditions — Coronary Disease; Dyslipidemias | interventions — 26S proteasome non-ATPase regulatory subunit 13

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Drug- Atorvastatin 40mg Dosage form- Oral tablet Frequency and duration- once daily for 28 days
  Interventions: Drug: Atorvo+™ (Arm1)
- Arm 2 (Experimental): Drug- Atorvo+™ Low (40 mg Atorvastatin and 100 mg CBD) Dosage form- Oral tablet Frequency and duration- once daily for 28 days
  Interventions: Drug: Atorvo+™ +CBD (Arm 2)
- Arm 3 (Experimental): Drug- Atorvo+™ High (40 mg Atorvastatin and 200 mg CBD) Dosage form- Oral tablet Frequency and duration- once daily for 28 days
  Interventions: Drug: Atorvo+™ +CBD (Arm 3)

INTERVENTIONS:
Drug: Atorvo+™ (Arm1) — Atorvo+™ is a combination product containing atorvastatin and cannabidiol (CBD).
  Arms: Arm 1
Drug: Atorvo+™ +CBD (Arm 2) — Atorvo+™ is a combination product containing atorvastatin and cannabidiol (CBD).
  Arms: Arm 2
Drug: Atorvo+™ +CBD (Arm 3) — Atorvo+™ is a combination product containing atorvastatin and cannabidiol (CBD).
  Arms: Arm 3

SUMMARY:
A Phase 1 study will assess the safety, tolerability, and pharmacokinetics of Atorvo+™ in healthy adult participants.

.

DETAILED DESCRIPTION:
This study will be testing an approved dose of atorvastatin (40 mg) and doses of CBD in the approved range (100 mg and 200 mg, approximately 1.7 mg/kg/day and 3.3 mg/kg/day for a 60 kg patient, respectively) in the study.

A total of 24 participants are planned to be enrolled into 3 study arms. Eight (8) participants are planned to be randomized in each of Arms 1, 2, and 3. Each arm will consist of a 28-days Screening period, a 28-day treatment period, and a 14-day follow-up period. Investigational products (IPs) refer to all study treatments and will be administered at the following planned dose levels:

* Arm 1: Atorvastatin (generic formulation) oral tablet 40 mg once daily for 28 days.
* Arm 2: Atorvo+™ Low (40 mg Atorvastatin and 100 mg CBD) once daily for 28 days.
* Arm 3: Atorvo+™ High (40 mg Atorvastatin and 200 mg CBD) once daily for 28 days.

ELIGIBILITY:
Diagnosis and Main Criteria for Inclusion:

Inclusion Criteria:

To be eligible for this study, a participant must meet all of the following inclusion criteria:

1. Able to and willing to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.
2. Male or female aged between 40 and 75 years (inclusive at the time of consent).
3. Nonsmoker (not used any tobacco products within 2 months prior to Screening). Participants who smoke ≤ 5 cigarettes or equivalent (eg, cigars, vaping, nicotine patches) per week can be included in the study at the discretion of the PI or designee if willing to abstain during inpatient stay.
4. Body mass index (BMI) >18.0 and <32.0 kg/m2 at Screening and body weight ≥50.0 kg and ≤ 120.0 kg.
5. Is judged by the Investigator to be in generally good health based on medical history, physical examination, vital sign parameters, ECG, laboratory parameters, and other relevant tests conducted at Screening.
6. Pulse between 50 and 100 beats per minute (bpm), inclusive at Screening.
7. Systolic blood pressure (BP) between 100 and 140 mmHg, diastolic BP between 50 and 90 mmHg inclusive, at Screening. For the purpose of qualifying any given participant for study participation, out-of-range vital signs may be repeated once.
8. No known allergic reaction to cannabis products (including tetrahydrocannabinol [THC], CBD, marijuana, and hashish) or EPIDIOLEX®.
9. Must have hepatic and renal clinical laboratory test results (total bilirubin and estimated glomerular filtrate rate [eGFR] by the CKD-EPI [2021] equation) within a laboratory defined normal range at Screening. Repeat testing at Screening is acceptable for out-of-range values following approval by the PI or designers.
10. Females must not be pregnant, lactating, or planning pregnancy, and if they are a woman of childbearing potential (WOCBP), must use acceptable, highly effective contraception from Screening until 93 days (90 days + approximately 5 half-lives) after the last IP administration. Effective forms of contraception are defined in Section 7.2.2. Females with same-sex partners (abstinence from penile-vaginal intercourse) are eligible when this is their preferred and usual lifestyle. Women of childbearing potential must have a negative serum hCG pregnancy test at Screening and negative urine test on Day -1. Women not of childbearing potential must be postmenopausal for ≥ 12 months (postmenopausal status is to be confirmed through testing of follicle-stimulating hormone [FSH] levels ≥ 40 IU/L at Screening for amenorrhoeic female participants), or otherwise permanently sterile (for which acceptable methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy).
11. Male participants who are sexually active with WOCBP must meet any of the following criteria:

    1. Vasectomy for at least 6 months prior to enrolment and willing and able to use a condom.
    2. Willing and able to use one of highly effective contraception methods.
    3. Male participants with pregnant partners are not eligible.
12. Male participants must be willing not to donate sperm throughout the study and for 93 days (90 days + approximately 5 half-lives) after the last dose of IP.
13. Willing and able to adhere to all study requirements, including willingness to remain in the study unit for the entire duration of the confinement period.
14. Participant has a good venous access bilaterally.

Exclusion Criteria:

A participant who meets any of the following exclusion criteria must be excluded from the study:

1. History of any clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine (including type 2 diabetes), oncologic, pulmonary, immunologic, or cardiovascular disease or other condition which could jeopardize safety or impact validity of results at the discretion of the PI.
2. Has any documented clinically significant infection, injury, or illness within 1 month prior to Screening.
3. Has any documented history of, or currently active, seizure disorder or history of clinically significant head injury.
4. Has an active malignancy of any type or has been diagnosed with cancer within 5 years prior to Screening (excluding squamous or basal cell carcinoma of the skin).
5. Any laboratory test results deemed clinically significant by the PI (clinically significant results may be repeated once at discretion of the investigator) or positive test for hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at Screening.
6. Positive COVID-19 polymerase chain reaction (PCR) test results at Day -1.
7. History of inherent cardiac abnormalities at the discretion of the PI.
8. Clinically significant ECG abnormalities (Fridericia's corrected QT interval [QTcF] >450 msec for males and >470 msec for females), PR >210 msec, QRS interval >120 msec at Screening (clinically significant results may be repeated once at discretion of the investigator).
9. ALT, AST, total cholesterol, LDL-C, or triglycerides >1.5 × the upper limit of normal (ULN) at Screening. Repeat testing at Screening is acceptable for out-of-range values following approval by the PI or designees.
10. Known allergic reactions to any excipient in the IP formulations.
11. History of significant drug abuse such as cocaine, phencyclidine (PCP), crack, opioid derivatives including heroin, and amphetamine derivatives within 1 year prior to Screening.
12. Use of marijuana or THC (directly or indirectly) within 90 days prior to drug administration and during the course of the study.
13. Positive screen for urine drug, urine cotinine (Day -1 only), or breath alcohol test at Screening or Day -1 (positive results may be repeated once at discretion of the investigator).
14. History of significant alcohol abuse within 1 year prior to Screening or regular use of alcohol within 6 months prior to Screening that exceeds 14 units of alcohol per week (1 unit = 150 mL of wine, 375 mL of mid strength beer, or 30 mL of 40% distilled alcohol).
15. Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or participant safety (eg, topical drug products without significant systemic absorption):

    1. Prescription medications (except for contraceptives) within 14 days prior to the first dose until end of the study;
    2. Monoamine oxidase inhibitors (MAOIs) within 28 days prior to dosing and during the study;
    3. Over-the-counter products and natural health products (including herbal remedies such as St. John's wort, homeopathic and traditional medicines), and antacid preparations within 14 days prior to the first dose up to end of study. Vitamins used as nutritional supplements in non-therapeutic doses may be accepted at the discretion of the PI or designee, but they must be stopped at least 48 hours before dosing and during the study.
    4. Any drugs known to induce or inhibit hepatic and renal drug metabolism within 30 days prior to the first dose and during the study.
    5. Any known CYP2C9 and CYP3A4 enzymes altering drugs (eg, amiodarone, fluconazole, ketoconazole, itraconazole, clarithromycin, ritonavir, erythromycin, etc.) within 28 days prior to the first dose and during the study.
    6. Any drug that has a significant impact on the central nervous system (CNS) including benzodiazepines (eg, diazepam, alprazolam, lorazepam), antipsychotic medications (eg, haloperidol, risperidone, quetiapine), antidepressants (eg, sertraline, fluoxetine, escitalopram), antiepileptic drugs (eg, phenytoin, carbamazepine, valproate) or sedative-hypnotics (eg, zolpidem, zopiclone, eszopiclone) within 30 days prior to the first dose and during the study.
    7. Any BP regularizing drugs including antihypertensive agents (eg, amlodipine, lisinopril, metoprolol), diuretics (eg, hydrochlorothiazide, furosemide, spironolactone), vasodilators (eg, hydralazine, nitroglycerin, minoxidil), alpha-blockers (eg, doxazosin, prazosin, terazosin) within 30 days prior to the first dose and during the study.
16. Consumption of beverages or foods that contain grapefruit or Seville oranges, or products containing these fruits, within 7 days prior to the first dose and during the study.
17. Use of any investigational or marketed drug or medical device in a clinical trial within 30 days of 5 half-lives (whichever is longer) prior to the first dose of IP administration, administration of a biological product in the context of a clinical research study within 90 days prior to IP administration, or concomitant participation in an investigational study involving no drug or device administration.
18. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 30 days prior to Day -1.
19. Participant is unwilling to refrain from strenuous exercise (including weightlifting) from 7 days prior to admission to the site until completion of the final Follow-up visit.
20. Any underlying physical or psychological medical condition that, in the opinion of the PI, could confound the results of the study or make it unlikely for the participant to comply with the protocol or complete the study per protocol.
21. Current suicidal ideation as assessed by the C-SSRS (Baseline/Screening) up to 1 month prior to Screening; Participants with a significant psychiatric history including previous suicide attempt or a lifetime history of suicidal ideation may be excluded at the discretion of the PI or designee.
22. Any reason which, in the opinion of the Investigator or Sponsor, would prevent the participant from participating in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and relationship of adverse events (AEs) | Baseline to End of study (Day 42) from first IP dose
Incidence of serious adverse events (SAEs) | Baseline to End of study (Day 42) from first IP dose
Incidence of adverse events of special interest (AESIs) | Baseline to End of study (Day 42) from first IP dose
  This includes clinically significant abnormal values in liver function tests (LFTs) (aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin), myopathy, myositis, myalgia, and type 2 diabetes
Number of participants with changes in laboratory parameters | Baseline to End of study (Day 42) from first IP dose
  hematology, biochemistry, coagulation, and urinalysis), physical examination, vital signs (blood pressure [BP], heart rate [HR], respiratory rate [RR], and body temperature), electrocardiogram (ECG) parameters.

SECONDARY OUTCOMES:
Changes in Columbia-Suicide Severity Rating Scale (C-SSRS score) | Baseline to End of study (Day 42) from first IP dose
PK Parameters- Maximum Plasma concentration (Cmax) | Baseline to End of study (Day 42) from first IP dose
PK Parameters- Time for maximum concentration (Tmax) | Baseline to End of study (Day 42) from first IP dose
PK Parameters- Area under Curve | Baseline to End of study (Day 42) from first IP dose
  Area under curve to the last measurable concentration (AUC0-t), Area under the curve of concentration versus time from zero to infinity (AUC0-∞) and %AUC extra will be assessed.
PK parameters-Elimination rate constant (Kel) | Baseline to End of study (Day 42) from first IP dose
PK parameters- Half-life (t½) | Baseline to End of study (Day 42) from first IP dose
To evaluate mitochondrial oxidative stress in Atorvo+™ vs atorvastatin. | Baseline to End of study (Day 42) from first IP dose
  This is measured by mean change in oxygen consumption rate (OCR) in Atorvo+ ™ vs atorvastatin (Baseline to EOS visit). Key parameters to be assessed- Basal respiration
To evaluate mitochondrial oxidative stress in Atorvo+™ vs atorvastatin. | Baseline to End of study (Day 42) from first IP dose
  This is measured by mean change in oxygen consumption rate (OCR) in Atorvo+ ™ vs atorvastatin (Baseline to EOS visit). Key parameters to be assessed- ATP production.
To evaluate mitochondrial oxidative stress in Atorvo+™ vs atorvastatin. | Baseline to End of study (Day 42) from first IP dose
  This is measured by mean change in oxygen consumption rate (OCR) in Atorvo+ ™ vs atorvastatin (Baseline to EOS visit). Key parameters to be assessed- Proton leak
To evaluate mitochondrial oxidative stress in Atorvo+™ vs atorvastatin. | Baseline to End of study (Day 42) from first IP dose
  This is measured by mean change in oxygen consumption rate (OCR) in Atorvo+ ™ vs atorvastatin (Baseline to EOS visit). Key parameters to be assessed- Maximal respiration.
To evaluate mitochondrial oxidative stress in Atorvo+™ vs atorvastatin. | Baseline to End of study (Day 42) from first IP dose
  This is measured by mean change in oxygen consumption rate (OCR) in Atorvo+ ™ vs atorvastatin (Baseline to EOS visit). Key parameters to be assessed- Reserve capacity.
To evaluate mitochondrial oxidative stress in Atorvo+™ vs atorvastatin. | Baseline to End of study (Day 42) from first IP dose
  This is measured by mean change in oxygen consumption rate (OCR) in Atorvo+ ™ vs atorvastatin (Baseline to EOS visit). Key parameters to be assessed-Non-mitochondrial respiration.

CONTACTS AND LOCATIONS:
Overall Officials: James E Smeeding, Study Chair — President, Indication Biosciences
Locations (1):
- Nucleus Network, Melbourne, Australia